CLINICAL TRIAL: NCT06850363
Title: ExaStim Upper Limb Home Use Clinical Validation Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Niche Biomedical, Inc. dba ANEUVO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EXA2504
Record Dates: First submitted 2025-02-04; First posted 2025-02-27 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Cervical Spinal Cord Injury
Keywords: Neuromodulation; Spinal Cord Therapy; Rehabilitation; Electrical Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcutaneous Spinal Stimulation in the home setting (Experimental): Subjects will perform activities of daily living in conjunction with the ExaStim over a 4-week period in the home setting. In each session, subjects will receive stimulation while performing therapist-prescribed activities of daily living. Stimulation must be utilized for a maximum of 300 -minutes per week and a minimum of 125-minutes per week. The time spent using stimulation during home sessions, and the number of sessions that patients perform each week, is flexible and is intended to facilitate the use of ExaStim within each participant's daily routine.
  Interventions: Device: ExaStim Stimulation System

INTERVENTIONS:
Device: ExaStim Stimulation System — Transcutaneous Spinal Cord Stimulation
  Other Names: ExaStim

SUMMARY:
This is a multi-center, observational, single-arm, 6-week home study to evaluate the safety and efficacy of transcutaneous spinal cord stimulation via the ExaStim system for 4 consecutive weeks used in the home setting for individuals with traumatic spinal cord injury. The study consists of a baseline evaluation and 1-week training period (Week 0), a 4-week stimulation period (Weeks 1-4), and a follow-up visit (Week 5), for a total expected duration of participation for each subject of six weeks.

DETAILED DESCRIPTION:
During the first week of the study, baseline measurements will be recorded for each subject and all eligible subjects and their caregivers will participate in a 1-week "Training Phase." Subsequently, subjects will perform activities of daily living and/or home exercises in conjunction with the ExaStim over a 4-week period in the home setting. In each session, subjects will receive stimulation while performing therapist-prescribed home exercises or activities of daily living. Stimulation must be utilized for a maximum of 300 -minutes per week and a minimum of 125-minutes per week. The time spent using stimulation during home sessions, and the number of sessions that patients perform each week, is flexible and is intended to facilitate the use of ExaStim within each participant's daily routine. Subjects and Clinicians will participate in weekly telehealth check-ins throughout the 4-week period in the home setting and will return to the clinic within one week of the final treatment to complete the final assessments in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have completed the ASPIRE clinical trial.
2. Subject must be ≥ 22 years of age at the time of the screening examination
3. Subject must have a traumatic, chronic* spinal cord injury between C2 and T2 inclusive
4. Subject must have American Spinal Injury Association (ASIA) Impairment Scale A, B, C, or D via the ISNCSCI exam
5. Subject must have limited function of upper extremities with ISNCSCI Upper Extremity Motor Score for each arm from 5 to 20 inclusive
6. Subject must have a non-zero score in least one of the UEMS C7, C8 and T1 muscles on either side
7. Subject must have regular availability of a caregiver and/or family member to assist with donning and doffing the device and to assist with completion of session-related report forms
8. Subject, caregiver, and/or family member must be available for all in-clinic study visits and adhere to the study protocol
9. Subject, caregiver and/or family member must be able to use a digital mobile device, have reliable access to internet, and be able to complete all study related forms and questionnaires
10. Subject and caregiver must be able to commit to participating in a six-week study, be willing to comply with study instructions, agree to make all office and telehealth appointments, engage in a minimum of 12-minutes of home activities with stimulation per week, and complete the entire course of the study
11. Subject must be a primary/fluent English speaker
12. Subject must be able and willing to read, comprehend and give Authorization for Use/Disclosure of Health Information (HIPAA) and informed consent

Exclusion Criteria:

1. Active implanted medical device for electrical stimulation
2. Other internal metallic objects of unknown or foreign origin (unidentifiable surgical implants, shrapnel, bullet fragments, etc.)
3. Botox injections to the upper limb in prior 6 months
4. Uncontrolled autonomic dysreflexia or orthostatic hypotension
5. BMI > 40.0 (morbid obesity)
6. Acute medical conditions under active treatment that would contraindicate standard rehabilitation including open wounds, unhealed bone fractures, peripheral neuropathies or painful musculoskeletal dysfunction
7. Subjects who are pregnant or planned pregnancy during the study. Note: Subjects of childbearing potential must agree to the use an effective contraceptive for the duration of the study.
8. Allergy to hydrogel, silicone, latex or other product materials
9. Compromised skin in the area for electrode contact (back of neck and/or hip area)
10. Uncontrolled cardiopulmonary disease
11. Ventilator dependency
12. Uncontrolled epilepsy or seizures
13. Unmanaged depression, psychiatric disorders or ongoing substance abuse
14. Participation in another clinical trial that may interfere with this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of device related adverse events | Occurrence over 6-weeks
  Incidence of device related adverse events over the course of the trial. no scoring requirement

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | change from baseline to week-5
  is an individualized, client-centered instrument designed to measure an individual's self-perception of physical functioning and satisfaction in the activities identified as important by the client. COPM score ranges from 0-50, higher scores mean a better outcome.
Patient Global Impression of Change (PGIC) | score at week 5
  The Patient Global Impression of Change Questionnaire is rated on a 10-point scale depicting a patient's rating of overall improvement. This self-reported scale reflects a patient's belief about the efficacy of treatment. score range from 0-10 with lower scores showing considerable imrpovement.
Psychosocial Impact of Assistive Devices Scale | score at week 5
  The PIADS Questionnaire is a 26-item self-reported questionnaire designed to assess the effects of an assistive device on functional independence, well-being and quality of life. Score range of 0-182 points with higher scores reflecting positive impact.
Capabilities of Upper Extremity Test | maintenance or change from baseline to week 5
  The CUE-T is an objective performance measure to assess upper extremity functional limitations in spinal cord injury individuals. CUE-T score ranges from 0 to 140, higher scores mean a better outcome.
Upper Extremity Motor Score | maintenance or change from baseline to week 5
  UEMS is a sub score of the ISNSCSCI. The ISNCSCI exam is a standardized tool traditionally used in clinical trials to broadly assess motor and sensory changes in individuals after spinal cord injury. The UEMS, a sub score of the ISNCSCI exam, better reflects meaningful recovery in the arms and hands, an area of utmost importance to individuals living with tetraplegia. The UEMS grades on a scale of 0-50, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Craig Rehabilitation Hospital, Denver, Colorado
  - TryAbility Neurorecovery Center, Downer Grove, Illinois
  - Internation Center for Spinal Cord Injury at the Kennedy Krieger Institute, Baltimore, Maryland
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Marquette University Neuro Recovery Clinic, Milwaukee, Wisconsin